CLINICAL TRIAL: NCT07191392
Title: Intervention Effect of Temporal Interference Stimulation (TIS) on Depressive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yanghua Tian, Vice President of Anhui Medical University, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AHMU-TIS-MDD
Record Dates: First submitted 2025-09-10; First posted 2025-09-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depressive Disorder; Temporal Interference Stimulation
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active TIS 10 to 14 times.
  Interventions: Device: Temporal Interference Stimulation (TIS)
- sham stimulation (Sham Comparator): Participants will receive sham TIS 10 to 14 times.
  Interventions: Device: Sham temporal interference stimulation (TIS)

INTERVENTIONS:
Device: Temporal Interference Stimulation (TIS) — The total stimulation duration was 30 minutes, including a 30-second current ramp-up at the beginning and a 30-second ramp-down at the end.
  Arms: real stimulation
Device: Sham temporal interference stimulation (TIS) — Sham stimulation had only 30 seconds of current ramping-up and ramping-down at the beginning and end of the stimulation, respectively, to simulate the sensation of actual stimulation
  Arms: sham stimulation

SUMMARY:
To investigate the effect of Temporal Interference Stimulation (TIS) on associative memory (AM) in patients with depressive disorder

DETAILED DESCRIPTION:
Depression group: thirty patients with depressive disorder diagnosed by DSM-5 were recruited from the Second Affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving TIS treatment. After meeting the inclusion criteria and obtaining informed consent. Each patient received either 30-minute or sham TIS.

Before and after the treatments, the patients had received a battery measure of neuropsychological tests, and MRI scan in multimodalities. Neuropsychological assessment included HAMD, ANSAQ, HAMA, PHQ15, BSSI, PSQI, ISI, RRS, Barratt,Buss&Perry and PVAQ. Multimodal MRI includes 3D-T1, rs-fMRI, and DTI.

Healthy controls: thirty healthy participants, who met the same exclusion criteria as the depressed patients but without a diagnosis of depression, were matched to the patients in terms of age, sex, and years of schooling.

The incidental memory task with emotional pictures were applied to evaluate the associative memory (AM) of thirty depressed patients at pre- and post-TIS compared to thirty healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for depression, and HAMD>17, BSS>6, PHQ-15>5.
* the age ranged from 18 to 65 years old, and the length of education was more than 5 years.
* the visual acuity or corrected visual acuity is normal, right-handed, can cooperate with the completion of various experimental tests.

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.
* accompanied by other neurological diseases, such as stroke, epilepsy and so on. pregnant and lactating women.
* accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
face-word assciative memory task score | baseline and immediately after the intervention
  In the face-cued word association test, participants viewed 12 grayscale photographs of faces on a computer screen, each shown for 4 seconds. Each photograph was paired with a distinct word, which participants read aloud when shown. Participants were instructed to memorize the word linked to each face. One minute later, participants viewed the same 12 faces in a new random order. They were then asked to recall the associated words. Each face was scored as correct or incorrect, and the total number of correct responses formed the AM score.
Change in Hamilton Depression Rating Scale (HAMD) Score | baseline and immediately after the intervention
  The HAMD is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
Change in the Patient Health Questionnaire-15 (PHQ-15) scale | baseline and immediately after the intervention
  The PHQ-15 is a 15-item scale to measure the severity of somatic symptoms, where each item is rated on a scale from 0 to 2. The PHQ-15 total score ranges from 0 to 30, with lower scores indicating less somatic symptoms.

SECONDARY OUTCOMES:
MRI measures | baseline and immediately after the intervention
  the functional connectivity between stimulated target and the whole brain areas; the global and regional activity measures.
Dot-probe Task | baseline and immediately after the intervention
  Using the Chinese Affective Face Picture System, select 20 negative emotional faces, 20 positive emotional faces, and 40 neutral emotional faces, with an equal ratio of male and female faces. Match the positive and negative faces with neutral faces respectively. Run a standardized dot-probe paradigm using E-Prime software.
  First, a fixation point is displayed in the center of the screen for 1000 ms, followed by a pair of face images for 1000 ms-one emotional face and one neutral face. After the images disappear, a probe will randomly appear on either the left or right side. Press "A" for the left side and "L" for the right side. Record the participants' reaction time and accuracy in response to positive-neutral, neutral-neutral, and negative-neutral image pairs to evaluate attentional bias. Shorter reaction times and higher accuracy indicate higher scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China